CLINICAL TRIAL: NCT05320575
Title: Zanubrutinib Monotherapy in Patients With Hemophagocytic Lymphohistiocytosis
Brief Title: Zanubrutinib for HLH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Principal Investigator, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Zanubrutinib HLH
Record Dates: First submitted 2022-04-02; First posted 2022-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: HLH
MeSH Terms: interventions — zanubrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- zanubrutinib (Experimental)
  Interventions: Drug: Zanubrutinib

INTERVENTIONS:
Drug: Zanubrutinib — The dosage of zanubrutinib is 160mg twice a day (80mg twice a day for patients over 75 years old) for 2 months. The remission rate is evaluated after treatment. If it is above PR, continue the dose maintenance treatment.

SUMMARY:
This study is a prospective single-arm clinical study, focusing on Hemophagocytic lymphohistocytosis，to evaluate the clinical efficacy and safety of zanubrutinib.

ELIGIBILITY:
Inclusion Criteria:

1. Unlimited gender, age ≥ 14 years old;
2. HLH was diagnosed according to HLH-04 diagnostic criteria;
3. Before the study, there was no severe liver function injury; Serum creatinine ≤ 1.5 times the upper limit of normal value;
4. Sign informed consent

Exclusion Criteria:

1. Allergic to zebutinib;
2. Currently active important cardiovascular diseases with clinical significance; The functions of important organs such as heart and lung unrelated to HLH were seriously abnormal;
3. Known human immunodeficiency virus (HIV) or active hepatitis B (HBV) or hepatitis C (HCV) infection;
4. Pregnant or lactating women and patients of childbearing age who refuse to take appropriate contraceptive measures during this trial;
5. Serious mental illness;
6. Active massive hemorrhage of internal organs;
7. Uncontrollable infection;
8. At the same time, participate in other clinical researchers

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
evaluation of treatment response | Change from before and 2,4,6 and 8 weeks after initiating therapy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT).
  A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5×109/L; for patients with a neutrophil count of 0.5 to 2.0× 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L,response was defined as an ALT decrease of at least 50%.
Progression Free Survival | 6 months
  from date of inclusion to date of progression, relapse, or death from any cause
Adverse events | 6 months
  Adverse events including myelosuppression, infection, hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China